CLINICAL TRIAL: NCT03693430
Title: Two-year Effect and Safety of Semaglutide 2.4 mg Once-weekly in Subjects With Overweight or Obesity
Brief Title: Two-year Research Study Investigating How Well Semaglutide Works in People Suffering From Overweight or Obesity
Acronym: STEP 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4378; 2017-003726-32 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1202-1740 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants will receive semaglutide 2.4 mg during 104-week treatment period in addition to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive placebo (semaglutide) during 104-week treatment period in addition to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: Placebo (Semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Subcutaneous (s.c., under the skin) injections of semaglutide once weekly at escalating doses (0.25 mg/week, 0.5 mg/week, 1.0 mg/week, 1.7 mg/week, 2.4 mg/week). The dose will be escalated to next level every 4 weeks
  Arms: Semaglutide
Drug: Placebo (Semaglutide) — S.c. injections of placebo once weekly at a similar dose escalation manner as semaglutide (placebo matched to semaglutide 0.25 mg/week, 0.5 mg/week, 1.0 mg/week, 1.7 mg/week, 2.4 mg/week). The dose will be escalated to next level every 4 weeks
  Arms: Placebo

SUMMARY:
This study will look at the change in body weight from the start to the end of the study. Researchers will compare the weight loss in people taking semaglutide (a new medicine) to people taking "dummy" medicine. In addition to taking the medicine, participants will also have talks with study staff about healthy food choices, how the participant can be more physically active and what participants can do to lose weight. Participants will either get semaglutide or "dummy" medicine - which treatment the participant gets is decided by chance. Participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm. The study will last for about 2 years. The participants will have 19 clinic visits and 15 phone calls with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age more than or equal to 18 years at the time of signing informed consent
* Body mass index (BMI) more than or equal to 30 kg/m^2 or more than or equal to 27 kg/m^2 with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease
* History of at least one self-reported unsuccessful dietary effort to lose body weight

Exclusion criteria:

* HbA1c more than or equal to 48 mmol/mol (6.5%) as measured by the central laboratory at screening
* A self-reported change in body weight more than 5 kg (11 lbs) within 90 days before screening irrespective of medical records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (37):
- United States (15):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Arlington, Virginia
- Canada (7):
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Moncton, New Brunswick
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Québec
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Komárom
  - Novo Nordisk Investigational Site, Szekszárd
- Italy (5):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Pisa
  - Novo Nordisk Investigational Site, Rome
  - Novo Nordisk Investigational Site, Siena
- Spain (6):
  - Novo Nordisk Investigational Site, Alcorcón
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, L'Hospitalet de Llobregat
  - Novo Nordisk Investigational Site, Pamplona
  - Novo Nordisk Investigational Site, Pozuelo de Alarcón
  - Novo Nordisk Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Kushner RF, Calanna S, Davies M, Dicker D, Garvey WT, Goldman B, Lingvay I, Thomsen M, Wadden TA, Wharton S, Wilding JPH, Rubino D. Semaglutide 2.4 mg for the Treatment of Obesity: Key Elements of the STEP Trials 1 to 5. Obesity (Silver Spring). 2020 Jun;28(6):1050-1061. doi: 10.1002/oby.22794. PMID 32441473
- [Background] Wharton S, Batterham RL, Bhatta M, Buscemi S, Christensen LN, Frias JP, Jodar E, Kandler K, Rigas G, Wadden TA, Garvey WT. Two-year effect of semaglutide 2.4 mg on control of eating in adults with overweight/obesity: STEP 5. Obesity (Silver Spring). 2023 Mar;31(3):703-715. doi: 10.1002/oby.23673. Epub 2023 Jan 18. PMID 36655300
- [Derived] Wadden TA, Brown GK, Egebjerg C, Frenkel O, Goldman B, Kushner RF, McGowan B, Overvad M, Fink-Jensen A. Psychiatric Safety of Semaglutide for Weight Management in People Without Known Major Psychopathology: Post Hoc Analysis of the STEP 1, 2, 3, and 5 Trials. JAMA Intern Med. 2024 Nov 1;184(11):1290-1300. doi: 10.1001/jamainternmed.2024.4346. PMID 39226070
- [Derived] Wilkinson L, Holst-Hansen T, Laursen PN, Rinnov AR, Batterham RL, Garvey WT. Effect of semaglutide 2.4 mg once weekly on 10-year type 2 diabetes risk in adults with overweight or obesity. Obesity (Silver Spring). 2023 Sep;31(9):2249-2259. doi: 10.1002/oby.23842. PMID 37605636
- [Derived] Garvey WT, Batterham RL, Bhatta M, Buscemi S, Christensen LN, Frias JP, Jodar E, Kandler K, Rigas G, Wadden TA, Wharton S; STEP 5 Study Group. Two-year effects of semaglutide in adults with overweight or obesity: the STEP 5 trial. Nat Med. 2022 Oct;28(10):2083-2091. doi: 10.1038/s41591-022-02026-4. Epub 2022 Oct 10. PMID 36216945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 41 sites in 5 countries as follows: Canada (9 sites), Hungary (6 sites), Italy (5 sites), Spain (6 sites), and United States (15 sites).
Pre-assignment Details: Participants were randomized in a 1:1 manner to receive treatment with semaglutide 2.4 milligram (mg) or placebo once weekly as an adjunct to a reduced-calorie diet and increased physical activity. The trial has a 104 weeks treatment period (16 weeks of dose escalation period and 88 weeks of maintenance dose).
Groups:
- Semaglutide 2.4 mg: Participants received once-weekly subcutaneous (s.c) injection of semaglutide in 16 week dose escalation period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg and 1.7 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached. Treatment was continued on the maintenance dose of 2.4 mg once weekly for an additional 88 weeks until week 104.
- Placebo: Participants received once-weekly s.c. injection of placebo matched to semaglutide for 104 weeks.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 152 | 152
Full Analysis Set (FAS) | 152 | 152
Safety Analysis Set (SAS) | 152 | 152
Completed | 148 | 134
Not Completed | 4 | 18
Not completed — Lost to Follow-up | 3 | 14
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised participants according to the intention-to-treat principle.
Groups:
- Semaglutide 2.4 mg: Participants received once-weekly s.c injection of semaglutide in 16 week dose escalation period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg and 1.7 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached. Treatment was continued on the maintenance dose of 2.4 mg once weekly for an additional 88 weeks until week 104.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 152 | 152 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12) | 47 (10) | 47 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 113 | 236
  Male | 29 | 39 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 21 | 39
  Not Hispanic or Latino | 134 | 131 | 265
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 141 | 142 | 283
  Black or African American | 7 | 5 | 12
  Other | 0 | 4 | 4
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline (Week 0) to Week 104 in Body Weight
Description: Percentage change in body weight for both in-trial and on-treatment observation period from baseline (week 0) to week 104 is presented. The outcome measure was evaluated based on the data from both in-trial and on-treatment periods. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site. On-treatment observation period: the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: From Baseline (Week 0) to Week 104
Population: The FAS included all randomised participants according to the intention-to-treat principle. Overall Number of Participants Analyzed = participants with available data for this outcome measure and Number Analyzed = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 144 | 128
percentage change
  In-trial observation period | -15.9 (12.3) | -1.9 (8.9)
  On-treatment observation period: number analyzed (Participants) | 132 | 109
  On-treatment observation period | -17.3 (11.9) | -2.0 (8.6)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority — Week 104 responses were analysed using an analysis of covariance model with randomised treatment as factor and baseline body weight as covariate. Missing observations were multiple (x1000) imputed from retrieved subjects of the same randomised treatment arm; p < .0001, ANCOVA; Treatment difference = -12.55, 95% CI 2-sided [-15.33 to -9.77]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Hypothetical estimand; Test type: Superiority — All responses prior to first discontinuation of treatment (or initiation of other anti-obesity medication or bariatric surgery) were included in a mixed model for repeated measurements with randomised treatment as factor and baseline body weight as covariate, all nested within visit; p < 0.0001, MMRM (Mixed model repeated measurement); Treatment difference = -16.05, 95% CI 2-sided [-18.64 to -13.45]

2. Primary Outcome: Number of Participants Who Achieved (Yes/no): Body Weight Reduction More Than or Equal to 5%
Description: Number of participants who achieved greater than or equal to (>=) 5% weight loss at 104 weeks is presented. In the reported data, 'Yes' infers the number of participants who have achieved >=5% weight loss, whereas 'No' infers the number of participants who have not achieved >=5% weight loss. The outcome measure was evaluated based on the data from both in-trial and on-treatment periods. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site. On-treatment observation period: the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: At Week 104
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 144 | 128
Participants
  In-trial observation period: Yes | 111 | 44
  In-trial observation period: No | 33 | 84
  On-treatment observation period: number analyzed (Participants) | 132 | 109
  On-treatment observation period: Yes | 110 | 38
  On-treatment observation period: No | 22 | 71
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.99, 95% CI 2-sided [2.95 to 8.42]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Hypothetical estimand; Test type: Superiority; p < 0.0001, MMRM; Odds Ratio (OR) = 18.06, 95% CI 2-sided [10.04 to 32.49]

3. Secondary Outcome: Number of Participants Who Achieved (Yes/no): Body Weight Reduction More Than or Equal to 10%
Description: Number of participants who achieved >=10% weight loss at 104 weeks is presented. In the reported data, 'Yes' infers the number of participants who have achieved >=10% weight loss, whereas 'No' infers the number of participants who have not achieved >=10% weight loss. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: At Week 104
Population: The FAS included all randomised participants according to the intention-to-treat principle. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 144 | 128
Participants
  Yes | 89 | 17
  No | 55 | 111

4. Secondary Outcome: Number of Participants Who Achieved (Yes/no): Body Weight Reduction More Than or Equal to 15%
Description: Number of participants who achieved >=15% weight loss at 104 weeks is presented. In the reported data, 'Yes' infers the number of participants who have achieved >=15% weight loss, whereas 'No' infers the number of participants who have not achieved >=15% weight loss. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: At Week 104
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 144 | 128
Participants
  Yes | 75 | 9
  No | 69 | 119

5. Secondary Outcome: Number of Participants Who Achieved (Yes/no): Body Weight Reduction More Than or Equal to 20%
Description: Number of participants who achieved >=20% weight loss at 104 weeks is presented. In the reported data, 'Yes' infers the number of participants who have achieved >=20% weight loss, whereas 'No' infers the number of participants who have not achieved >=20% weight loss. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: At Week 104
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 144 | 128
Participants
  Yes | 52 | 3
  No | 92 | 125

6. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to week 104 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 143 | 126
centimeter (cm) | -15.2 (12.4) | -4.3 (9.1)

7. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Body Weight (kg)
Description: Change in body weight from baseline (week 0) to week 104 in kilogram (kg) is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 144 | 128
kilogram | -16.9 (14.0) | -2.1 (9.5)

8. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Body Mass Index (BMI)
Description: Change in BMI from baseline (week 0) to week 104 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 144 | 128
kilogram per square meter (kg/m^2) | -6.2 (5.3) | -0.7 (3.5)

9. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline (week 0) to week 104 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 142 | 125
millimeter of mercury (mmHg) | -6 (13) | -1 (15)

10. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from baseline (week 0) to week 104 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 142 | 125
mmHg | -4 (10) | -1 (9)

11. Secondary Outcome: Change in Total Cholesterol-ratio to Baseline
Description: Change in total cholesterol from baseline (week 0) to week 104 measured in milligrams per deciliter (mg/dL) is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 141 | 121
Ratio of total cholesterol | 0.96 (15.3) | 1.02 (13.5)

12. Secondary Outcome: Change in High Density Lipoprotein (HDL) Cholesterol-ratio to Baseline
Description: Change in HDL cholesterol from baseline (week 0) to week 104 measured in mg/dL is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 141 | 120
Ratio of HDL cholesterol | 1.09 (19.1) | 1.08 (15.4)

13. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol-ratio to Baseline
Description: Change in LDL cholesterol from baseline (week 0) to week 104 measured in mg/dL is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 141 | 121
Ratio of LDL cholesterol | 0.93 (23.8) | 0.99 (19.1)

14. Secondary Outcome: Change in Very Low Density Lipoprotein (VLDL) Cholesterol-ratio to Baseline
Description: Change in VLDL cholesterol from baseline (week 0) to week 104 measured in mg/dL is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 141 | 121
Ratio of VLDL cholesterol | 0.79 (42.3) | 1.03 (35.1)

15. Secondary Outcome: Change in Free Fatty Acids-ratio to Baseline
Description: Change in free fatty acids from baseline (week 0) to week 104 measured in mg/dL is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 133 | 111
Ratio of free fatty acids | 0.99 (71.2) | 1.07 (69.1)

16. Secondary Outcome: Change in Triglycerides-ratio to Baseline
Description: Change in triglycerides from baseline (week 0) to week 104 measured in mg/dL is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 141 | 121
Ratio of triglycerides | 0.79 (42.4) | 1.03 (36.0)

17. Secondary Outcome: Change in High Sensitivity C-reactive Protein (hsCRP)-Ratio to Baseline
Description: Change in hsCRP from baseline (week 0) to week 104 measured in mg/dL is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of hsCRP
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 141 | 121
Ratio of hsCRP | 0.41 (149.1) | 0.99 (105.5)

18. Secondary Outcome: Change in Glycated Haemoglobin (HbA1c) (Percent [%])
Description: Change in HbA1c from baseline (week 0) to week 104 in % is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent of glycated haemoglobin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 141 | 122
Percent of glycated haemoglobin | -0.5 (0.3) | -0.1 (0.3)

19. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in HbA1c (mmol/Mol)
Description: Change in HbA1c from baseline (week 0) to week 104 in millimole per mole (mmol/mol) is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 141 | 122
mmol/mol | -5.1 (3.2) | -1.0 (3.0)

20. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Fasting Plasma Glucose (FPG) (mmol/L)
Description: Change in FPG from baseline (week 0) to week 104 in millimoles per liter (mmol/L) is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 137 | 117
mmol/L | -0.5 (0.5) | 0.1 (0.6)

21. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in FPG (mg/dL)
Description: Change in FPG from baseline (week 0) to week 104 in mg/dL is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 137 | 117
mg/dL | -8.3 (9.6) | 1.8 (10.8)

22. Secondary Outcome: Change in Fasting Serum Insulin-ratio to Baseline (Pmol/L)
Description: Change in fasting serum insulin from baseline (week 0) to week 104 measured in picomole per liter (pmol) is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting serum insulin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 110
Ratio of fasting serum insulin | 0.68 (54.1) | 0.96 (62.9)

23. Secondary Outcome: Change in Fasting Serum Insulin-ratio to Baseline (mIU/mL)
Description: Change in fasting serum insulin from baseline (week 0) to week 104 measured in milli-international units per milliliter (mIU/mL) is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting serum insulin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 110
Ratio of fasting serum insulin | 0.68 (54.1) | 0.96 (62.9)

24. Secondary Outcome: Percentage Change From Baseline (Week 0) to Week 52 in Body Weight
Description: Percentage change in body weight from baseline (week 0) to week 52 is presented.
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 149 | 129
percentage change | -15.8 (9.3) | -3.3 (6.4)

25. Secondary Outcome: Change From Baseline (Week 0) to Week 52 in Body Weight (kg)
Description: Change in body weight from baseline (week 0) to week 52 in kg is presented.
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 149 | 129
kilogram (kg) | -16.7 (10.3) | -3.5 (7.4)

26. Secondary Outcome: Change From Baseline (Week 0) to Week 52 in Body Mass Index (BMI)
Description: Change in BMI from baseline (week 0) to week 52 is presented.
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 149 | 129
kilogram per square meter (kg/m^2) | -6.1 (3.8) | -1.3 (2.6)

27. Secondary Outcome: Change From Baseline (Week 0) to Week 52 in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to week 52 is presented.
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 149 | 129
centimeter (cm) | -14.3 (9.4) | -4.5 (6.8)

28. Secondary Outcome: Number of Participants Who at 52 Weeks Achieved (Yes/no): Body Weight Reduction More Than or Equal to 5%
Description: Number of participants who achieved >=5% weight loss at 52 weeks is presented. In the reported data, 'Yes' infers the number of participants who have achieved >=5% weight loss, whereas 'No' infers the number of participants who have not achieved >=5% weight loss.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 149 | 129
Participants
  Yes | 132 | 38
  No | 17 | 91

29. Secondary Outcome: Number of Participants Who at 52 Weeks Achieved (Yes/no): Body Weight Reduction More Than or Equal to 10%
Description: Number of participants who achieved >=10% weight loss at 52 weeks is presented. In the reported data, 'Yes' infers the number of participants who have achieved >=10% weight loss, whereas 'No' infers the number of participants who have not achieved >=10% weight loss.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 149 | 129
Participants
  Yes | 102 | 17
  No | 47 | 112

30. Secondary Outcome: Number of Participants Who at 52 Weeks Achieved (Yes/no): Body Weight Reduction More Than or Equal to 15%
Description: Number of participants who achieved >=15% weight loss at 52 weeks is presented. In the reported data, 'Yes' infers the number of participants who have achieved >=15% weight loss, whereas 'No' infers the number of participants who have not achieved >=15% weight loss.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 149 | 129
Participants
  Yes | 78 | 7
  No | 71 | 122

31. Secondary Outcome: Number of Participants Who at 52 Weeks Achieved (Yes/no): Body Weight Reduction More Than or Equal to 20%
Description: Number of participants who achieved >=20% weight loss at 52 weeks is presented. In the reported data, 'Yes' infers the number of participants who have achieved >=20% weight loss, whereas 'No' infers the number of participants who have not achieved >=20% weight loss.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 149 | 129
Participants
  Yes | 52 | 3
  No | 97 | 126

32. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned here are TEAE defined as an event that had onset date (or increase in severity) on or after the first day of exposure to treatment. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from first to last trial product administration plus 7 weeks of follow-up and excluding any period of temporary treatment interruption defined as >7 consecutive missed doses (corresponding to >7 weeks off-treatment).
Time Frame: From Baseline (Week 0) to Week 111
Population: The safety analysis set (SAS) included all randomised participants exposed to at least one dose of randomised treatment.
Measure: Number; unit: events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 152 | 152
events | 1645 | 1059

33. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: A SAE was defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. The SAEs occurred from week 0 to week 111 is presented. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from first to last trial product administration plus 7 weeks of follow-up and excluding any period of temporary treatment interruption defined as >7 consecutive missed doses (corresponding to >7 weeks off-treatment).
Time Frame: From Baseline (Week 0) to Week 111
Population: The SAS included all randomised participants exposed to at least one dose of randomised treatment.
Measure: Number; unit: events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 152 | 152
events | 18 | 20

34. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Pulse
Description: Change in pulse from baseline (week 0) to week 104 is presented. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: From Baseline (Week 0) to Week 104
Population: The SAS included all randomised participants exposed to at least one dose of randomised treatment. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 130 | 106
beats per minute (beats/min) | 3 (10) | -1 (9)

35. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Amylase
Description: Change in amylase from baseline (week 0) to week 104 is presented. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Units/liter (U/L)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 130 | 106
Units/liter (U/L) | 1.13 (20.7) | 1.02 (15.1)

36. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Lipase
Description: Change in lipase from baseline (week 0) to week 104 is presented. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 130 | 106
U/L | 1.47 (52.3) | 1.00 (34.4)

37. Secondary Outcome: Change From Baseline (Week 0) to Week 104 in Calcitonin
Description: Change in calcitonin from baseline (week 0) to week 104 is presented. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per liter (ng/L)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 124 | 102
nanogram per liter (ng/L) | 0.99 (21.5) | 0.97 (41.0)

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0) to Week 111
Description: All AEs mentioned here are TEAE defined as an event that had onset date (or increase in severity) on or after the first day of exposure to randomized treatment and no later than the date of last dose + 7 weeks. Results are based on the SAS which included all randomized participants exposed to at least one dose of randomized treatment.
Arm/Group | Semaglutide 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/152 | 0/152
Serious Adverse Events (participants affected / at risk) | 12/152 | 18/152
Other Adverse Events (participants affected / at risk) | 141/152 | 117/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=152) | Placebo (N=152)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=152) | Placebo (N=152)
Abdominal distension (Gastrointestinal disorders) | 15 (22) | 9 (13)
Abdominal pain (Gastrointestinal disorders) | 20 (32) | 4 (14)
Abdominal pain upper (Gastrointestinal disorders) | 22 (23) | 10 (13)
Anxiety (Psychiatric disorders) | 8 (8) | 11 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (20) | 11 (20)
Asthenia (General disorders) | 8 (10) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 19 (20)
Bronchitis (Infections and infestations) | 8 (9) | 8 (9)
COVID-19 (Infections and infestations) | 15 (16) | 6 (6)
Constipation (Gastrointestinal disorders) | 47 (62) | 17 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (10)
Decreased appetite (Metabolism and nutrition disorders) | 17 (18) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 53 (108) | 36 (51)
Dizziness (Nervous system disorders) | 13 (16) | 8 (12)
Dyspepsia (Gastrointestinal disorders) | 20 (24) | 7 (12)
Eructation (Gastrointestinal disorders) | 17 (21) | 1 (2)
Fatigue (General disorders) | 11 (12) | 8 (8)
Flatulence (Gastrointestinal disorders) | 20 (25) | 10 (11)
Gastroenteritis (Infections and infestations) | 20 (28) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (19) | 6 (6)
Headache (Nervous system disorders) | 16 (36) | 16 (31)
Hypertension (Vascular disorders) | 6 (6) | 14 (14)
Influenza (Infections and infestations) | 20 (23) | 16 (19)
Injection site bruising (General disorders) | 5 (8) | 8 (11)
Ligament sprain (Injury, poisoning and procedural complications) | 10 (10) | 1 (1)
Nasopharyngitis (Infections and infestations) | 24 (33) | 23 (31)
Nausea (Gastrointestinal disorders) | 81 (213) | 33 (53)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 8 (9)
Sinusitis (Infections and infestations) | 8 (8) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 20 (31) | 23 (30)
Urinary tract infection (Infections and infestations) | 12 (19) | 6 (7)
Vomiting (Gastrointestinal disorders) | 46 (78) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT03693430/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT03693430/SAP_001.pdf